CLINICAL TRIAL: NCT01075503
Title: New Approach for Brachial Plexus Block: Clinical Research of Retrograde Infraclavicular Brachial Plexus Blockade
Brief Title: Clinical Research of Retrograde Infraclavicular Brachial Plexus Blockade
Acronym: RIBPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Xin Youqing, Beijing jishuitan hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: JSTMZ.1
Record Dates: First submitted 2010-02-22; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Upper Extremity
Keywords: Supraclavicular; Interscalene; Infraclavicular; Brachial plexus block; Ropivacaine
MeSH Terms: interventions — Brachial Plexus Block

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- retrograde infraclavicular (Experimental): Patients were received retrograde infraclavicular brachial plexus block.
  Interventions: Procedure: brachial plexus block
- interscalene (Active Comparator): Patients were received interscalene brachial plexus block.
  Interventions: Procedure: brachial plexus block
- supraclavicular (Active Comparator): Patients were received supraclavicular brachial plexus block.
  Interventions: Procedure: brachial plexus block

INTERVENTIONS:
Procedure: brachial plexus block — 0.5% Ropivacaine 40ml
  Other Names: NAROPIN® 1.0%

SUMMARY:
Brachial plexus block is a frequently used technique for upper extremity surgery. All present approaches and techniques have certain advantages and disadvantages. It's necessary to develop a new approach to brachial plexus block which 1) provides reliable anesthesia, 2) is easy to perform, 3) isn't restricted by posture, 4) provides extensive sensory distribution, 5) causes as few complications as possible, 6) easily place a secured catheter for post-operative analgesia. The investigators established the retrograde infraclavicular brachial plexus block approach. The investigators compared and verified the feasibility, efficacy and safety of this new approach with other classic approaches to brachial plexus block.

DETAILED DESCRIPTION:
Traditional brachial plexus block approaches have certain limitations. This study evaluated the effectiveness, safety and feasibility of a new retrograde infraclavicular brachial plexus block as compared with interscalene and supraclavicular approaches. 90 patients scheduled for elective upper limb surgery were recruited and randomized into three groups, 30 for each group. Patients of Group A received retrograde infraclavicular block, interscalene (by Winnie) approach for Group B and supraclavicular (by Kulenkampff) approach for Group C. The retrograde infraclavicular block was performed with the insertion point medial to the coracoid process and the needle advanced to ipsilateral interscalene groove. Neurostimulation was used and 40ml of 0.5% ropivacaine were injected. Sensory block, adverse effects and complications were evaluated and recorded every 5 minutes until 30min after local anesthetic injection. The needle insertion depth, angles in coronary and sagittal planes of Group A were also recorded. Success rate of each nerve sensory block, sensory block result, complications, rate of satisfaction, rate of failure and incidence rate of adverse effects are all compared among groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status Ⅰ~Ⅱ
* Scheduled for elective upper extremity surgery

Exclusion Criteria:

* Age <18 yr or >60 yr
* Body weight <50kg or >100kg
* Serious brain, heart, lung, liver, kidney diseases or diabetes mellitus
* Incapability or refusing to be enrolled
* Infection at the site of puncture, skin ulcer
* Coagulopathy
* Contralateral phrenic nerve paralysis, contralateral recurrent laryngeal nerve paralysis or pneumothorax

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Success rate of nerve sensory block | 30 minutes

SECONDARY OUTCOMES:
Success rate of motor block | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoguang Zhang, MB, Principal Investigator — Department of anesthesiology, Beijing jishuitan hospital, China
Locations (1):
- Beijing jishuitan hospital, Beijing, China